CLINICAL TRIAL: NCT06348121
Title: Efficacy of Bifidobacterium Animalis Subsp. Lactis and Lacticaseibacillus Rhamnosus Mixture in Children With ADHD
Brief Title: Impact of Probiotics on Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WK2024003
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic group (Experimental): 5B CFU/strip/day WecProB, before meal
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of the study had last 56 days, and each patient will make 3 visits (d0, d28, d56).

SUMMARY:
This study investigates WecProB (Bifidobacterium animalis subsp. lactis and Lacticaseibacillus rhamnosus) to evaluate their potential to improve symptoms and safety in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ADHD per DSM-5 criteria;
2. Age 6-12 years, gender-neutral;
3. IQ >70 on intelligence testing;
4. Participant/guardian comprehension and voluntary consent.

Exclusion Criteria:

1. Those with a clear history of other serious neurological diseases, such as epilepsy, head trauma, encephalitis or meningitis, etc.;
2. Have taken antibiotics, probiotics or immunosuppressants within one month before starting the experiment;
3. Ongoing special diet, such as ketogenic diet, etc
4. BMI higher than the 90th percentile or lower than the 10th percentile for children of the same age and sex;
5. Those who have had symptoms of respiratory or digestive tract infection in the past month, such as fever, cough, diarrhea, etc.;
6. Those who have had inflammatory bowel disease in the past, such as ulcerative colitis, Crohn's disease, etc.;

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms of ADHD | 56 days
  The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2), was employed to assess the executive functioning deficits commonly associated with ADHD in children. The BRIEF-2 scale ranges from a minimum of 0 to a maximum of 300 points. Higher scores on the BRIEF-2 indicate greater executive dysfunction, meaning that a higher score reflects worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Niu Q, Wang W, Liang Y, Fang S, Wan L, Yang G. Efficacy and Safety of a Probiotic Mixture Containing Bifidobacterium animalis subsp. lactis BLa80 and Lacticaseibacillus rhamnosus LRa05 in Children With Attention-Deficit/Hyperactivity Disorder. Mol Nutr Food Res. 2025 Nov;69(22):e70234. doi: 10.1002/mnfr.70234. Epub 2025 Sep 2. PMID 40898729